CLINICAL TRIAL: NCT04130594
Title: Double-blind, Placebo-controlled Study With an Open Dose Selection Period for Assessing the Safety and Immunogenicity of the Drug "BVRS-GamVac", a Vector Vaccine for the Prevention of the Middle East Respiratory Syndrome, Lyophilisate for the Preparation of a Solution for Intramuscular Administration, With the Participation of Healthy Volunteers
Brief Title: Study of Safety and Immunogenicity of BVRS-GamVac
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01-BVRS-GamVac-2019
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: MERS (Middle East Respiratory Syndrome); MERS
Keywords: vaccine; vector based vaccine; Middle East respiratory syndrome; Immunologic Factors; Physiological Effects of Drugs; MERS-Cov
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: This clinical trial is designed as a double blind randomized placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- phase 1, vaccine half dose (Experimental): half dose of BVRS-GamVac vaccine single administration
  Interventions: Biological: BVRS-GamVac
- phase 1, vaccine full dose (Experimental): full dose of BVRS-GamVac vaccine single administration
  Interventions: Biological: BVRS-GamVac
- phase 2, vaccine selected dose (Experimental): selected dose of BVRS-GamVac vaccine single administration
  Interventions: Biological: BVRS-GamVac
- phase 2, placebo (Placebo Comparator): placebo single administration
  Interventions: Other: placebo

INTERVENTIONS:
Biological: BVRS-GamVac — a vector vaccine for the prevention of the Middle East respiratory syndrome, lyophilisate for the preparation of a solution for intramuscular administration
  Arms: phase 1, vaccine full dose; phase 1, vaccine half dose; phase 2, vaccine selected dose
Other: placebo — placebo
  Arms: phase 2, placebo

SUMMARY:
The Middle East respiratory syndrome coronavirus (MERS-CoV) was identified in 2012 during the first Middle East respiratory syndrome (MERS) outbreak. MERS-CoV causes an acute lower-respiratory infection in humans, with a fatality rate of ~34.5%.

The aim of the study is to assess the safety and immunogenicity of adenoviral-based vaccine against MERS - BVRS-GamVac.

DETAILED DESCRIPTION:
Two-stage, open-dose, prospective, double-blind, randomized, placebo-controlled study in parallel groups The study will include volunteers of both sexes, aged 18-55 years inclusive. The study will involve 162 (will receive the study drug or placebo) healthy volunteers, of which the first stage, it is planned to vaccinate 40 person with the studied drug (at the same time, the participation of 8 spares *), at the second phase - 122 people, of whom 88 will receive the study drug, and 34 will make up the control group of observation - they will be given a placebo drug.

* Volunteers are replaced by spares before the introduction of the drug, if the volunteer took the drug, then its replacement is not performed.

Any volunteer who received a dose of the test drug will be considered as included in the study, the data available on it will be used in assessing the safety and tolerability of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent;
2. absence of a history, as well as according to a screening examination of pathology from the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, urogenital, immune and endocrine systems, blood, which may affect volunteer safety and evaluation of the results of the study (clinical, instrumental and laboratory studies did not reveal diseases or clinically significant deviations);
3. males and females within the age range from 18 to 55 years;
4. Consent to the use of effective methods of contraception during the entire period of participation in the study;
5. subject body mass index (BMI): 18.5 ≤ BMI ≤ 30;
6. absence of acute infectious diseases at the time of vaccination and 7 days before vaccination;
7. absence of severe allergic diseases in the medical history
8. no serious post-vaccination complications in patient's history following the earlier administration of immunobiological products;
9. subject has a negative result of the blood or urine pregnancy test (for females of childbearing age);
10. subject has negative tests for HIV, hepatitis B and С, syphilis;
11. subject has a negative result of the urine test for residual narcotic drugs;
12. Negative alcohol test;
13. The indicators of the complete blood count test and biochemical analysis of blood on the screen within 1,1*ULN/LLN (upper limit of normal/lower limit of normal)
14. absence of inflammatory or dystrophic myocardial changes based on ECG data

Exclusion Criteria:

1. Volunteer participation in any other study over the past 90 days;
2. Any vaccination in the last 30 days;
3. Acute infectious and non-infectious diseases, exacerbations of chronic diseases within 4 weeks prior to screening;
4. subject has received treatment with steroids for the last 10 days;
5. subject has received immunoglobulins or other blood products over the last 3 months;
6. subject has received immunosuppressive and/or immunomodulating agents within 6 months prior to the start of the study;
7. Pregnancy or lactation;
8. subject has systolic blood pressure less than 100 mm Hg or greater than 139 mm Hg; diastolic blood pressure less than 60 mm Hg or greater than 90 mm Hg; heart rate lower than 60 beats per minute or above 100 beats per minute;
9. A burdened allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, a history of serum sickness, hypersensitivity or allergic reactions to the introduction of any vaccines in history, known allergic reactions to vaccine components, etc.);
10. Diabetes mellitus or other forms of impaired glucose tolerance;
11. presence of a concomitant illness in decompensation stage which might affect the course of the study (CNS organic lesion, decompensated cardiovascular diseases, any manifestations of kidney or acute liver failure, oncological diseases, diabetes mellitus);
12. subject has a a history of neoplasms (ICD codes C00-D09);
13. blood donation (at least 450 ml of blood or plasma) by subject in less than 2 months prior to the start of the study;
14. Reception of narcotic and psychostimulating drugs at present or in the anamnesis;
15. subject has a history of the consumption of more than 5 units alcohol per week, alcohol intake within 48 hours before the injection of the test drug;
16. subject smokes more than 10 cigarettes a day;
17. subject has a planned hospitalization and / or surgery during the period of participation in the study, as well as 4 weeks before the estimated date of vaccination.
18. subject has any condition that, according to the researcher's doctor, may be a contraindication to participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | through the whole study, an average of 180 days
  Determination of Number of Participants With Adverse Events
Number of Participants With Serious Adverse Events | through the whole study, an average of 180 days
  Determination of Number of Participants With Serious Adverse Events
Number of Participants with Solicited Local and Systemic Adverse Events | through the whole study, an average of 180 days
  Determination of Number of Participants with Solicited Local and Systemic Adverse Events
Antibody levels against the MERS-CoV glycoprotein S measured by an enzyme-linked immunosorbent assay (ELISA) | at days 0, 7, 14, 21, 28, 42, 56 and 90
  Determination of antibody levels against the MERS-CoV glycoprotein S measured by an ELISA vs. baseline values (phase 1, phase 2) and placebo (phase 2)

SECONDARY OUTCOMES:
Assessment of antigen-specific cell-mediated immune response | at 0 and 14 days from the start of vaccination compared to baseline values (day 0)
  determination of specific T-cell- mediated response vs. baseline values (phase 1, phase 2) and placebo (phase 2)
Neutralizing antibody levels | at days 0, 14 and 28
  Determination of the neutralizing antibody titer for a virus in virus neutralization reaction vs. baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No